CLINICAL TRIAL: NCT04903119
Title: A Phase 1 Study of Nilotinib in Combination With Dabrafenib and Trametinib or Encorafenib/Binimetinib in BRAF V600 Mutant Metastatic Melanoma After Progression on BRAF/MEK Inhibition
Brief Title: Nilotinib Plus Dabrafenib/Trametinib or Encorafenib/Binimetinib in Metastatic Melanoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ruta Arays (Other)
Collaborators: Novartis (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Ruta Arays, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20-MEL-11-PMC; 1R01CA258751-01A1 (NIH)
Record Dates: First submitted 2021-04-26; First posted 2021-05-26 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Melanoma; BRAF Gene Mutation
Keywords: dose escalation; nilotinib; dabrafenib; trametinib; pharmacokinetics; CYP3A4; encorafenib; binimetinib
MeSH Terms: conditions — Melanoma | interventions — nilotinib; dabrafenib; trametinib; encorafenib; binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Level 1 (Experimental): Patients in this group will receive 100mg Nilotinib PO BID.
  Interventions: Drug: Nilotinib 100mg; Drug: Dabrafenib; Drug: Trametinib; Drug: Encorafenib; Drug: Binimetinib
- Level 2 (Experimental): Patients in this group will receive 200mg Nilotinib PO BID.
  Interventions: Drug: Nilotinib 200mg; Drug: Dabrafenib; Drug: Trametinib; Drug: Encorafenib; Drug: Binimetinib
- Level 3 (Experimental): Patients in this group will receive 300mg Nilotinib PO BID.
  Interventions: Drug: Nilotinib 300mg; Drug: Dabrafenib; Drug: Trametinib; Drug: Encorafenib; Drug: Binimetinib
- Level 4 (Experimental): Patients in this group will receive 400mg Nilotinib PO BID.
  Interventions: Drug: Nilotinib 400mg; Drug: Dabrafenib; Drug: Trametinib; Drug: Encorafenib; Drug: Binimetinib

INTERVENTIONS:
Drug: Nilotinib 100mg — Patients will begin dabrafenib (150mg PO BID) and trametinib (2mg PO once daily) or encorafenib (450 mg PO) and binimetinib (45 mg PO BID) on day one and will continue for 28 days. After 7 days, nilotinib will be added at 100mg PO BID and will continue for 21 days. For each subsequent cycle, nilotinib will be given for 28 days.
  Arms: Level 1
Drug: Nilotinib 200mg — Patients will begin dabrafenib (150mg PO BID) and trametinib (2mg PO once daily) or encorafenib (450 mg PO) and binimetinib (45 mg PO BID) on day one and will continue for 28 days. After 7 days, nilotinib will be added at 200mg PO BID and will continue for 21 days. For each subsequent cycle, nilotinib will be given for 28 days.
  Arms: Level 2
Drug: Nilotinib 300mg — Patients will begin dabrafenib (150mg PO BID) and trametinib (2mg PO once daily) or encorafenib (450 mg PO) and binimetinib (45 mg PO BID) on day one and will continue for 28 days. After 7 days, nilotinib will be added at 300mg PO BID and will continue for 21 days. For each subsequent cycle, nilotinib will be given for 28 days.
  Arms: Level 3
Drug: Nilotinib 400mg — Patients will begin dabrafenib (150mg PO BID) and trametinib (2mg PO once daily) or encorafenib (450 mg PO) and binimetinib (45 mg PO BID) on day one and will continue for 28 days. After 7 days, nilotinib will be added at 400mg PO BID and will continue for 21 days. For each subsequent cycle, nilotinib will be given for 28 days.
  Arms: Level 4
Drug: Dabrafenib — All patients will begin dabrafenib (150mg PO BID) on day one and will continue for 28 days.
Drug: Trametinib — All patients will begin trametinib (2mg PO once daily) on day one and will continue for 28 days.
Drug: Encorafenib — encorafenib will be administered orally 450mg once daily for 28 consecutive days
Drug: Binimetinib — binimetinib will be administered orally 45mg twice daily for 28 consecutive days

SUMMARY:
This is a phase 1 dose-escalation study of nilotinib in combination with fixed-dose dabrafenib and trametinib regimen for patients with metastatic or unresectable melanoma carrying a BRAF V600 mutation and have relapsed on a BRAF/MEK inhibitor therapy. The goal is to assess the toxicity and tolerability and determine the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of the combination of nilotinib with dabrafenib and trametinib or with encorafenib and binimetinib. Additionally, this study will assess pharmacokinetic parameters of dabrafenib and nilotinib when used in combination.

DETAILED DESCRIPTION:
This is a phase 1 dose-escalation study of nilotinib in combination with a fixed-dose of dabrafenib and trametinib or with encorafenib and binimetinib. The first week, patients will be treated with dabrafenib (150mg, twice daily) and trametinib (2mg, once daily), or encorafenib (450 mg, daily) and binimetinib (45 mg twice daily). After 7 days, when both drugs have achieved steady-state levels and there is maximal induction of CYP3A4, nilotinib will be added, and all three drugs dosed concurrently for the rest of the study. Plasma pharmacokinetic (PKs) samples for dabrafenib and nilotinib will be obtained at baseline, weekly for the first four weeks, and at regular study visits for the duration of the trial. Tissue core biopsies and correlative plasma samples will be obtained at baseline, and 2 weeks after the start of nilotinib.

ELIGIBILITY:
Inclusion Criteria

* Patients must have histologically confirmed metastatic or unresectable melanoma. Radiological evaluation should occur within 28 days prior to enrollment initiation.
* Patients must have a BRAF V600 mutation. Any CLIA-certified mutation testing is acceptable to document mutation status.
* Patients must have stable disease on dabrafenib and trametinib or on encorafenib and binimetinib for a duration of greater than or equal to 3 months OR have failed any BRAFi/MEKi regimen to qualify for the trial, including the dabrafenib/trametinib combination and/or the encorafenib/ binimetinib combination.
* Patient may have had prior immunotherapy for metastatic disease or prior cellular therapy (although NOT mandatory). NOTE: Other prior therapies are not allowed, with the exception of radiation.
* Age ≥18 years.
* ECOG performance status ≤ 1.
* Patients must have adequate organ and marrow function as defined below:
* absolute neutrophil count ≥1,500/mcL
* platelets ≥100,000/mcL
* total bilirubin ≤ institutional upper limit of normal (ULN)
* AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
* creatinine ≤ institutional ULN OR
* glomerular filtration rate (GFR) ≥60 mL/min/1.73 m2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m2.
* Patients with known human immunodeficiency virus (HIV) on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with known history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a known history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with known HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with treated brain metastases are eligible if follow-up brain imaging 4 weeks or longer after central nervous system (CNS)-directed therapy shows no evidence of progression.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* Measurable (target) disease by Response Evaluation Criteria In Solid Tumors (RECIST 1.1) criteria. Target lesions selected for tumor measurements should be those where additional (e.g., palliative) treatments are not indicated or anticipated.

  • Measurable disease per RECIST 1.1 requirements: defined as longest diameter to be recorded for non-nodal lesions > 10mm and short axis for nodal lesions >15 mm using conventional techniques
* The effects of nilotinib, encorafenib, dabrafenib, binimetinib and trametinib on the developing human fetus are unknown, women of childbearing potential and men must agree to use adequate contraception (non-hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of nilotinib, dabrafenib, and trametinib administration.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Patients with chronic hypokalemia or chronic hypomagnesemia. Patients can be eligible with a repeat screening, if results show repletion.
* Patients with long QT syndrome or baseline QTc (Fridericia) >470 msec in males and >480 msec in females (ULN for each respectively).
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1 or greater than baseline) with the exception of alopecia, grade 2 fatigue, vitiligo or endocrinopathies on stable replacement therapy).
* Patients who are receiving any other investigational therapies that could affect the primary or secondary outcomes of this study.
* Untreated brain metastases are not allowed.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nilotinib, dabrafenib, encorafenib, binimetinib and trametinib.
* Patients receiving any medications or substances that are strong CYP3A inhibitors are ineligible for this trial. Patients receiving any medications or substances that are strong CYP3A inducers are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Patients receiving any medications or substances that are strong CYP2C8 inhibitors are ineligible for the dabrafenib+ trametinib. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Use of proton pump inhibitors concurrent with nilotinib is prohibited. Use of short-acting antacids or H2 blockers as an alternative to proton pump inhibitors is allowable.
* Use of drugs or substances known to prolong QT interval is prohibited with Nilotinib
* Patients with uncontrolled intercurrent illness.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or lactating women

Inclusion of Women and Minorities

-There are no exclusions for trial participation based on gender nor race.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients Experiencing Dose Limiting Toxicities | 28 days
  Percentage of patients who experienced dose-limiting toxicities associated with Nilotinib as defined by the study protocol.

SECONDARY OUTCOMES:
Dose-Adjusted Steady State Concentration of Dabrafenib | 15 days
  The dose-adjusted steady state concentrations (Css) of dabrafenib will be calculated on day 8 (dabrafenib alone) compared to day 15 (dabrafenib + nilotinib).
Change in Nilotinib Concentration | 1 month
  Plasma concentrations of Nilotinib will be measured on day 8 (pre-Nilotinib) and day 29.
Duration of Response | 12 months
  Duration of overall response will be determined by the time measurement criteria are met for complete response (CR) or partial response (PR) - whichever is first recorded - until the first date that recurrent or progressive disease is objectively documented.

CONTACTS AND LOCATIONS:
Overall Officials: Ruta Arays, MD, Principal Investigator — University of Kentucky
Locations (4):
- United States (4):
  - University of Iowa, Iowa City, Iowa
  - Markey Cancer Center, Lexington, Kentucky
  - St. Luke's University Health Network, Easton, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No